CLINICAL TRIAL: NCT01629693
Title: Clinical Evaluation of Two Monthly Replacement Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A00973
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Myopia; Astigmatism
Keywords: contact lenses; myopia; astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix (Experimental): Lotrafilcon B contact lenses worn bilaterally (in both eyes) for at least 4 hours a day, 5 days a week, for 4 weeks, on a daily wear basis (removed nightly for cleaning and disinfection).
  Interventions: Device: Lotrafilcon B contact lenses
- Biofinity (Active Comparator): Comfilcon A contact lenses worn bilaterally (in both eyes) for at least 4 hours a day, 5 days a week, for 4 weeks, on a daily wear basis (removed nightly for cleaning and disinfection).
  Interventions: Device: Comfilcon A contact lenses

INTERVENTIONS:
Device: Lotrafilcon B contact lenses — Silicone hydrogel contact lenses (sphere or toric) per subject's habitual prescription
  Other Names: AIR OPTIX® AQUA; AIR OPTIX® for ASTIGMATISM
  Arms: Air Optix
Device: Comfilcon A contact lenses — Silicone hydrogel contact lenses (sphere or toric) per subject's habitual prescription
  Other Names: Biofinity® Sphere; Biofinity® Toric
  Arms: Biofinity

SUMMARY:
The purpose of this study is to evaluate differences in the comfort at the end of the month between Air Optix® lenses versus Biofinity® lenses in habitual daily wear symptomatic soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Must sign written informed consent document.
* Currently wearing weekly/biweekly or monthly sphere or toric soft contact lenses (NOT including AIR OPTIX Aqua, AIR OPTIX NIGHT & DAY Aqua, AIR OPTIX for Astigmatism, Biofinity Sphere, Biofinity Toric, or ProClear Toric soft contact lenses) bilaterrally (in both eyes) and have worn these lenses for at least 3 months, daily wear use only (no extended wear).
* Symptomatic for contact lens-related ocular discomfort at the end of the lens wearing day.
* Current contact lens prescription within the available parameters of both study products.
* Able to achieve visual acuity (VA) of at least 6/7.5 (20/25) in each eye with study lenses in the available parameters.
* Willing to wear study lenses for at least 4 hours/day and at least 5 days/week for the 1 month trial period.
* Willing and able to follow instructions, study procedures and maintain the appointment schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Neophytes and current wearers of AIR OPTIX Aqua, AIR OPTIX NIGHT & DAY Aqua, AIR OPTIX for Astigmatism, Biofinity sphere, Biofinity Toric, or ProClear Toric soft contact lenses.
* Any systemic or ocular disease or disorder (refractive disorder allowed and dry eye is permitted), complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* Recent (within 7 days of enrollment) or current ocular infections, active ocular inflammation, glaucoma or preauricular lymphadenopathy.
* A history of ocular surgery/trauma within the last 6 months.
* Topical or systemic antibiotics use within 7 days of enrollment.
* Topical ocular or systemic corticosteroids use within 14 days of enrollment.
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, Ph.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 22 sites located in the United States.
Pre-assignment Details: Of the 398 enrolled, 17 participants were exited as screen failures. This reporting group includes all participants who provided informed consent, were randomized, and utilized the study lenses (381).
Groups:
- Air Optix; Biofinity: Contact lenses worn bilaterally for at least 4 hours a day, 5 days a week, for 4 weeks, on a daily wear basis
Period: Overall Study
Arm/Group | Air Optix | Biofinity
Started | 193 | 188
Completed | 188 | 178
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Investigator decision | 0 | 1
Not completed — Poor comfort of study lenses | 0 | 2
Not completed — Subject decision unrelated to AE | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants who utilized the study lenses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Optix | Biofinity | Total
Number analyzed (Participants) | 193 | 188 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.1) | 33.1 (10.5) | 32.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 131 | 274
  Male | 50 | 57 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Likert Response: "I Can Comfortably Wear my Lenses" at Day 30
Description: Overall comfort was assessed by the participant as a response to the questionnaire item 'I can comfortably wear my lenses', using a 10-point Likert scale, with 1=poor and 10=excellent.
Time Frame: Baseline, Day 30
Population: This analysis population includes all participants who completed the protocol and had no major protocol violations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Air Optix | Biofinity
Number analyzed (Participants) | 179 | 168
units on a scale
  Baseline | 6.1 (2.2) | 6.3 (2.1)
  Change from Baseline at Day 30 | 1.5 (2.8) | 1.4 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from 10 Jul 2013 to 20 Nov 2013. AEs were obtained through volunteered and elicited comments from the participants.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device. This analysis population includes all participants enrolled and exposed to test and control articles.
Arm/Group | Air Optix | Biofinity
Serious Adverse Events (participants affected / at risk) | 1/193 | 1/188
Other Adverse Events (participants affected / at risk) | 0/193 | 0/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Air Optix (N=193) | Biofinity (N=188)
Acanthamoeba keratitis (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.